CLINICAL TRIAL: NCT00431236
Title: A Phase III Multicenter, Randomized, Double-Blind, Active-Controlled, Parallel Group Study of the Efficacy and Safety of the Intravenous and Oral Formulations of the Neurokinin-1 Receptor Antagonist, Casopitant, Administered in Combination With ZOFRAN and Dexamethasone for Prevention of Chemotherapy-Induced Nausea and Vomiting in Cancer Subjects Receiving Highly Emetogenic Cisplatin-Based Chemotherapy
Brief Title: A Study of the Drug Casopitant for the Prevention of Nausea Caused By Cisplatin-Based Highly Emetogenic Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: NKV102551
Record Dates: First submitted 2007-02-02; First posted 2007-02-05 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Nausea and Vomiting, Chemotherapy-Induced
Keywords: cisplatin; CINV; highly emetogenic
MeSH Terms: conditions — Nausea; Vomiting | interventions — casopitant; Ondansetron; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Oral Casopitant (GW679769)
Drug: IV Casopitant (GW679769)
Drug: IV ondansetron hydrochloride
Drug: Oral dexamethasone
  Other Names: IV ondansetron hydrochloride; IV Casopitant (GW679769); Oral Casopitant (GW679769)

SUMMARY:
This is a Phase III trial designed to demonstrate that casopitant when added to dexamethasone and ondansetron is more effective in the prevention of vomiting then dexamethasone and ondansetron alone, in patients who receive a cisplatin-based highly emetogenic chemotherapy.

DETAILED DESCRIPTION:
A Phase III Multicenter, Randomized, Double-Blind, Active-Controlled, Parallel Group Study of the Efficacy and Safety of the Intravenous and Oral Formulations of the Neurokinin-1 Receptor Antagonist, Casopitant, administered in Combination with ZOFRAN and Dexamethasone for Prevention of Chemotherapy-Induced Nausea and Vomiting in Cancer Subjects Receiving Highly Emetogenic Cisplatin-Based Chemotherapy

ELIGIBILITY:
Inclusion criteria:

* Subject understands the nature and purpose of this study and the study procedures and has signed an informed consent form for this study to indicate this understanding.
* Males or females of at least 18 years of age.
* Diagnosed with a malignant solid tumor and is scheduled to receive their first course of cytotoxic chemotherapy with cisplatin administered as a single intravenous dose of ≥ 70mg/m² over 1-4 hours on study Day 1, either alone or in combination with other chemotherapeutic agents. For combination regimens, non-cisplatin agents of moderate to high emetogenic potential will be allowed, but must be administered following the cisplatin infusion and be completed no more than 6 hours after the initiation of the cisplatin infusion. Chemotherapy agents of minimal to low emetogenic potential may be given on Day 1 following cisplatin or on any subsequent study day. Taxanes (e.g. paclitaxel, docetaxel) may be administered on study Day 1 only following cisplatin.
* Has an ECOG Performance Status of 0, 1, or 2.
* Hematologic and metabolic status must be adequate for receiving a highly emetogenic cisplatin-based regimen and meet the following criteria:

  * Total Neutrophils ≥ 1500/mm³ (Standard units : ≥1.5 x 10^9/L)
  * Platelets ≥ 100,000/mm (Standard units: ≥100.0 x 10^9/L)
  * Bilirubin ≤ 1.5 x ULN
  * Serum Creatinine ≤1.5 mg/dL (Standard units : ≤ 132.6 µMOL/L OR
  * Creatinine clearance ≥ 60 mL/min

Creatinine clearance must be calculated using the Cockcroft-Gault formula:

Clcreat (ml/min) = (140-age [yr]) x body wt [kg] 72 x serum creatinine [mg/dl] For females: multiply creatinine clearance by a factor of 0.85. OR Clcreat (ml/min) = (140-age [yr]) x body wt [kg] serum creatinine [µmol/L] K=1.05 for females K=1.23 for males

* Liver enzymes must be below the following limits:
* Without known liver metastases: Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) ≤ 2.5 x upper limit of normal.
* With known liver metastases: AST and/or ALT ≤ 5.0 x upper limit of normal.

  * Is willing and able to complete daily components of the subject diary for each study cycle.
  * Women of childbearing potential; must commit to consistent and correct use of an acceptable method of birth control; GSK acceptable contraceptive methods, when used consistently and in accordance with both the product label and the instructions of a physician, are as follows:

    1. non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal. For purposes of this study, postmenopausal is defined as one year without menses)
    2. child-bearing potential: must have a negative serum pregnancy test result or negative urine dipstick pregnancy test within 24 hours prior to the first dose of investigational product of cycle 1 day 1, and agrees to one of the following:
* male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for that female subject oral contraceptives (e.g., oral, injectable, or implantable) with double-barrier method of contraception consisting of spermicide with either condom or diaphragm for a period after the trial to account for a potential drug interaction (minimum of six weeks)
* double-barrier method of contraception consisting of spermicide with either condom or diaphragm
* intra-uterine device (IUD) with a documented failure rate of less than 1% per year
* complete abstinence from intercourse for two weeks before exposure to the investigational product throughout the clinical trial, and for a period after the trial to account for elimination of the drug (minimum of three days)
* if subjects indicate they will remain abstinent during the period described above, they must agree to follow GSK guidelines for the consistent and correct use of an acceptable method of birth control should they become sexually active.

obstruction

Exclusion criteria:

* Has previously received cytotoxic chemotherapy. Previous biological or hormonal therapy will be permitted.
* Is scheduled to receive cisplatin treatment on more than one day during a single cycle of therapy.
* If female, is pregnant or lactating.
* Has received radiation therapy to the thorax, head & neck, abdomen, or the pelvis in the 10 days prior to receiving the first dose of study medication and/or will receive radiation therapy to the thorax, head & neck, abdomen or the pelvis in the 6 days following the first dose of study medication.
* Emesis (i.e. vomiting and/or retching) experienced in the 24 hours prior to receiving the first dose of study medication.
* Clinically significant nausea (e.g. ≥25 mm on a VAS) in the 24 hours prior to receiving the first dose of study medication.
* A known central nervous system primary or malignancy metastatic to the CNS, unless successfully treated with excision or radiation and subsequently has been stable for at least 1 week prior to receiving the first dose of study medication.
* Has history of documented peptic ulcer disease (via endoscopy or x-ray), active peptic ulcer disease, gastrointestinal obstruction, increased intracranial pressure, hypercalcemia, or any uncontrolled medical condition (other than malignancy) which in the opinion of the Investigator may confound the results of the study, represent another potential etiology for emesis and nausea (other than CINV) or pose an unwarranted risk to the subject.
* Has a known hypersensitivity or contraindication to ZOFRAN, another 5-HT3 receptor antagonist, dexamethasone, or any component of casopitant.
* Has previously received an NK-1 receptor antagonist.
* An active systemic infection or any uncontrolled disease (other than malignancy) which, in the opinion of the investigator, may confound the results of the study or pose an unwarranted risk to the subject. Subjects with a previous, but not current, history of alcoholism may be permitted provided that, in the investigator's opinion, the subject's disease state will not confound the results of the study.
* Receiving or planning to receive a systemic corticosteroid therapy at any dose within 72 hours prior to the first dose of study medication, except where indicated as premedication for a taxane. However, topical steroids and inhaled corticosteroids with a steroid dose of≤10 mg prednisone daily or its equivalent are permitted.
* Is scheduled to receive bone marrow transplantation and/or stem cell rescue with this course of cisplatin therapy.
* Has received an investigational drug within the 30 days or five half-lives (whichever is longer) prior to receiving the first dose of study medication, and/or is scheduled to receive any investigational drug during the study.
* Has received moderately and/or highly emetogenic medication within the 48 hours prior to the first dose of study medication. (Opioid narcotics for cancer pain will be permitted if the subject has been on such medication for at least 7 days and has not experienced nausea or emesis from the narcotics.)
* Has taken/received any medication with known or potential antiemetic activity within the 24-hour period prior to receiving study drug. This includes, but is not limited to:

  * 5-HT3 receptor antagonists (e.g., ondansetron, granisetron, dolasetron, tropisetron, ramosetron). Palonestron is not permitted within 7 days prior to administration of investigational product.
  * benzamide / benzamide derivatives (e.g., metoclopramide, alizapride)
  * benzodiazepines (except if the subject is receiving such medication for sleep or anxiety and has been on a stable dose for at least seven days prior to the first dose of GW679769 investigational product; however, lorazepam is prohibited 24 hours prior to receiving study drug regardless of reason for use.)
  * phenothiazines (e.g., prochlorperazine, promethazine, fluphenazine, perphenazine, thiethylperazine, chlorpromazine)
  * butyrophenone (e.g., haloperidol, droperidol)
  * corticosteroids (e.g., dexamethasone, methylprednisolone; with the exception of topical steroids for skin disorders, inhaled steroids for respiratory disorders, and prophylactic treatment for taxane or pemetrexed therapy)
  * anticholinergics (e.g., scopolamine with the exception of inhaled anticholingerics for respiratory disorders e.g., ipratropium bromide)
  * antihistamines (e.g., cyclizine, hydroxyzine, diphenhydramine), except for prophylactic use for taxane therapy
  * domperidone
  * mirtazapine
  * olanzapine
  * cannabinoids
* Has taken/received strong or moderate inhibitors of CYP3A4 and CYP3A5 prior to administration of casopitant (GW679769) investigational product
* Has taken/received inducers of CYP3A4 and CYP3A5 within fourteen days prior to the administration of casopitant investigational product
* Is taking the anti-diabetic agent repaglinide or the diuretic torsemide. Investigators are advised to exercise caution if including patients taking the anti-diabetic agents rosiglitazone or pioglitazone, or antimalarial agents such as chloroquine and amodiaquine, as the metabolite of casopitant is a potential inhibitor of CYP2C8
* Is currently taking or plans to take any of the following CYP3A4 substrates: astemizole, cisapride, pimozide, terfenadine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 810 (Actual)
Dates: Start 2006-11-06 (Actual); Primary Completion 2007-10-09 (Actual); Study Completion 2007-10-09 (Actual)

PRIMARY OUTCOMES:
Number of participants who achieved complete response | Up to 120 hours of cycle 1 of HEC
  Complete response was defined as no vomiting/retching and no rescue therapy) over the first 120 hours following the initiation of their first cycle of a cisplatin-based HEC regimen. Vomiting was defined as the forceful expulsion of gastrointestinal contents through the mouth or nose. Retching was defined as the labored, spasmodic, rhythmic contraction of the respiratory and abdominal muscles in an attempt to vomit, that was not productive of gastrointestinal contents (also known as "dry heaves").

SECONDARY OUTCOMES:
Number of participants who achieved complete response during the acute (0-24 hours) and the delayed (24-120 hours) phase following the first cycle of HEC | Up to 120 hours of cycle 1 of HEC
  Complete response was defined as no vomiting/retching and no rescue therapy over the first 120 hours following the initiation of their first cycle of a cisplatin-based HEC regimen. Vomiting was defined as the forceful expulsion of gastrointestinal contents through the mouth or nose. Retching was defined as the labored, spasmodic, rhythmic contraction of the respiratory and abdominal muscles in an attempt to vomit, that was not productive of gastrointestinal contents (also known as "dry heaves").
Number of participants who achieved a complete response during the overall (0-120 hours) phase following subsequent cycles of HEC | Up to 120 hours of cycle of HEC 2 to 6
  Complete response was defined as no vomiting/retching and no rescue therapy over the first 120 hours following the initiation of their first cycle of a cisplatin-based HEC regimen. Vomiting was defined as the forceful expulsion of gastrointestinal contents through the mouth or nose. Retching was defined as the labored, spasmodic, rhythmic contraction of the respiratory and abdominal muscles in an attempt to vomit, that was not productive of gastrointestinal contents (also known as "dry heaves").
Maximum nausea score (to assess the severity of nausea), as assessed by a visual analogue scale (VAS) | Up to 120 hours of each HEC cycle (up to 24 months)
  Nausea was defined as a subjectively unpleasant sensation associated with the awareness of the urge to vomit; the desire to vomit without the presence of expulsive muscular movements. The participants were asked to rate the level of nausea he/she has experienced over the previous 24 hours for a period of 120 hours on a 100-point VAS scale (millimeters [mm]) where, 0: no nausea and 100: nausea as bad as it could be. Higher score indicates more severity. The maximum nausea score (to assess the severity of nausea) was assessed by a VAS during the acute (0-24 hour), delayed (24-120 hour) and overall (0-120 hour) phase.
Number of participants who use of anti-emetic rescue medication | Up to 120 hours of each HEC cycle (up to 24 months)
  Anti-emetic rescue medication was defined as any medication, other than the protocol prescribed agents, given specifically for the treatment or prophylaxis of nausea and/or emesis during the 120 hour assessment phase of each study cycle. The time to the first anti-emetic rescue medication was defined as the length of time from initiation of HEC until the time of first use of anti-emetic rescue medication.
Number of participants with first emetic event | Up to 120 hours of each HEC cycle (up to 24 months)
  Vomiting was defined as the forceful expulsion of gastrointestinal contents through the mouth or nose and retching was defined as the labored, spasmodic, rhythmic contraction of the respiratory and abdominal muscles in an attempt to vomit, that is not productive of gastrointestinal contents (also known as "dry heaves"). The time to first emetic event was defined as the length of time from initiation of HEC until the time of the first emetic event (example: retch/vomiting).
Number of participants who received anti-emetic rescue medication | Up to 120 hours of cycle 1 of HEC
  Anti-emetic rescue medication was defined as any medication, other than the protocol prescribed agents, given specifically for the treatment or prophylaxis of nausea and/or emesis during the 120 hour assessment phase of each study cycle. The time to the first anti-emetic rescue medication was defined as the length of time from initiation of HEC until the time of first use of anti-emetic rescue medication. If no event had occurred at the end of the 120 hour time period, then the observation was censored for the purpose of this analysis.
Number of participants who vomited/retched | Up to 120 hours of cycle 1 of HEC
  The forceful expulsion of gastrointestinal contents through the mouth or nose. The laboured, spasmodic, rhythmic contraction of the respiratory and abdominal muscles in an attempt to vomit, that was not productive of gastrointestinal contents (also known as "dry heaves"). It was assessed during the acute (0-24 hour), delayed (24-120 hour) and overall (0-120 hour) phase. The odds ratio indicated a reduction in the likelihood of vomiting in the single dose oral group and in the 3-Day IV/oral group compared with the control group.
Number of participants who reported significant nausea (>=25 mm on the VAS) | Up to 120 hours of cycle 1 of HEC
  Nausea was defined as a subjectively unpleasant sensation associated with the awareness of the urge to vomit; the desire to vomit without the presence of expulsive muscular movements. The participants were asked to rate the level of nausea he/she has experienced over the previous 24 hours for a period of 120 hours on a 100-point VAS scale (mm) where, 0: no nausea and 100: nausea as bad as it could be. Higher score indicates more severity. The maximum nausea score (to assess the severity of nausea) was assessed by a VAS during the acute (0-24 hour), delayed (24-120 hour) and overall (0-120 hour) phase.
Number of participants who reported nausea (>=5 mm on the VAS) | Up to 120 hours of cycle 1 of HEC
  Nausea was defined as a subjectively unpleasant sensation associated with the awareness of the urge to vomit; the desire to vomit without the presence of expulsive muscular movements. The participants were asked to rate the level of nausea he/she has experienced over the previous 24 hours for a period of 120 hours on a 100-point VAS scale (mm) where, 0: no nausea and 100: nausea as bad as it could be. Higher score indicates more severity. The maximum nausea score (to assess the severity of nausea) was assessed by a VAS during the acute (0-24 hour), delayed (24-120 hour) and overall (0-120 hour) phase.
Number of participants who achieved complete protection, defined as no vomiting/retching, no significant nausea and no rescue medication | Up to 120 hours of cycle 1 of HEC
  Complete protection was defined as no vomiting/retching, no rescue therapy and no significant nausea (<25 mm on VAS). It was assessed during the acute (0-24 hour), delayed (24-120 hour) and overall (0-120 hour) phase.
Number of participants who achieved total control, defined as no vomiting/retching, no nausea and no rescue medication | Up to 120 hours of each HEC cycle (up to 24 months)
  Total control was defined as no vomiting, no retching, no rescue therapy and no nausea (<5 mm on VAS). It was assessed during the acute (0-24 hour), delayed (24-120 hour) and overall (0-120 hour) phase.
The impact on participants daily life activities for the first 120 hours following the first cycle of chemotherapy as assessed by the Functional Living Index-Emesis (FLIE) questionnaire-Score | Up to 120 hours of each HEC cycle (up to 24 months)
  The FLIE was a self-administered questionnaire consisting of 18 items indicating impact of nausea and vomiting on daily activities: physical, social and emotional function, and the ability to enjoy meals. Questions are divided into two domains: nausea 1-9; vomiting 10-18. Each item was scored on a VAS from 1: not at all to 7: a great deal; higher score indicates more severity. The initial score for each question was calculated by measuring the distance from the left hand end to the point where the participant had placed the mark. For questions 1, 2, 4, 5, 7-10, 12-14, 16 and 17, the final score: subtracting the initial score from 100 and for questions 3, 6, 11, 15 and 18, final score was the one provided in the dataset. The score for the nausea/vomiting domain was the sum of the individual scores divided by the number actually answered multiplied by 9. This sum was then multiplied by 0.06 and 9 added. The score ranged from 9-63 for each nausea and vomiting and sum both is provided.
Percentage of participants with impact on daily life activities for the first 120 hours following the first cycle of chemotherapy as assessed by the FLIE questionnaire-interpretation | Up to 120 hours of each HEC cycle (up to 24 months)
  The FLIE was a self-administered questionnaire consisting of 18 items indicating impact of nausea and vomiting on daily activities: physical, social and emotional function, and the ability to enjoy meals. Questions are divided into two domains: nausea questions 1-9; vomiting questions 10-18. Each item was scored on a VAS from 1: not at all to 7: a great deal. Higher scores indicate less impairment on daily life as a result of nausea or vomiting. No impact on daily life was defined as an average item score of >6 on the 7-point scale. The total score for no impact of chemotherapy induced nausea and vomiting (CINV) daily life, defined as a FLIE total score of >108 (range: 18-126). The same method was applied to vomiting and nausea subscores: no impact of vomiting (nausea) on daily life was defined as a FLIE total score of >54 (range: 9-63). The FLIE total score, as well as the vomiting and nausea subscores, for each treatment arm was calculated at Baseline and Day 6-10.
Participant satisfaction with the prophylactic anti-emetic regimens, as assessed by the participant satisfaction questionnaire | Up to 120 hours of each HEC cycle (up to 24 months)
  A participant satisfaction questionnaire was included in the participants diary card. At Day 6-10 of cycle 1, participants were asked to rate overall satisfaction with study medications in preventing chemotherapy induced nausea and vomiting, using the 5-point scale: 1: very satisfied; 2: somewhat satisfied; 3: neither satisfied nor dissatisfied; 4: somewhat dissatisfied and 5: very dissatisfied, where higher score indicates greater dissatisfaction.
The willingness of participant to use the same treatment during future chemotherapy, as assessed by the participant willingness questionnaire | Up to 120 hours of each HEC cycle (up to 24 months)
  A participant willingness questionnaire was included in the participants diary card. Participants completed this assessment on Day 6 - 10. Participants were asked to rate overall willingness to use study medications in preventing chemotherapy induced nausea and vomiting, using the 5-point scale: 1: definitely would be willing; 2: probably would be willing; 3: not certain; 4: probably would not be willing and 5: definitely would not be willing.
Number of participants with nausea as assessed by a categorical scale, over the first 120 hours following HEC | Up to 120 hours of each HEC cycle (up to 24 months)
  Nausea was defined as a subjectively unpleasant sensation associated with the awareness of the urge to vomit; the desire to vomit without the presence of expulsive muscular movements. The categorical scale assessed the participant's severity of his/her nausea using the descriptions; none: no nausea, mild: queasiness/upset stomach that was manageable and minimally (if at all) affects daily activities; moderate: increased queasiness, sometimes with the feeling of having to vomit/throw up (but not vomiting), that has significant negative effect on the daily activities (for example, being unable to work, eat and drink, prepare food, care for children or others) and severe: feeling sick and vomiting or feeling like you are going to vomit and unable to perform most daily activities.
Number of participants with adverse events (AE) and serious adverse events (SAE) | Up to 24 month after last dose of investigational product
  An AE was defined as any untoward medical occurrence (MO) in a participant temporally associated with the use of a medicinal product (MP), whether or not considered related to the MP and can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with its use. The SAE was any untoward MO that, at any dose, results in death, life threatening, persistent or significant disability/incapacity, results in or prolongs inpatient hospitalization, congenital abnormality or birth defect, that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition.
Number of participants with abnormalities of Grade 3 and 4 in laboratory parameters (clinical chemistry and hematology) | Up to end of cycle (approximately 28 days per cycle); maximum up to 24 months
  Grade shifts from Baseline were assessed as shift from any Grade to Grade 3 or Grade 4 in any cycle. Toxicities were graded according to the National Cancer Institute common toxicity criteria for adverse events (NCI-CTCAE), version 3.0. Grade refers to the severity of the toxicity. The NCI-CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each toxicity based on the following general guideline: Grade 1: Mild AE, Grade 2: Moderate AE, Grade 3: Severe AE, Grade 4: Life-threatening or disabling AE and Grade 5: Death related to AE. It was assessed on Day 1, during day 6-10 and end of cycle. Clinical chemistry parameters assessed included: alkaline phosphatase (ALP), alanine amino transferase (ALT), aspartate amino transferase (AST), total bilirubin, creatinine, blood urea nitrogen (BUN), chloride, glucose, potassium, sodium and urea. Hematology parameters assessed included: hemoglobin, hematocrit, total neutrophils, platelets and white blood cells (WBC).
Summary of abnormal electrocardiogram findings | Up to end of cycle (approximately 28 days per cycle); maximum up to 24 months
  It was assessed on Day 1, during day 6-10 and end of cycle. Electrocardiogram data clinically significant change from Baseline (worse, improved and no change) is presented.
Summary of mean systolic blood pressure (SBP) and diastolic blood pressure (DBP) | Up to end of cycle (approximately 28 days per cycle); maximum up to 24 months
  It was assessed on Day 1, during day 6-10 and end of cycle in cycle 1 while on Day 1 and end of cycle in subsequent cycles 2 to 6. Summary of mean SBP and DBP is presented.
Summary of mean respiratory rate | Up to end of cycle (approximately 28 days per cycle); maximum up to 24 months
  It was assessed on Day 1, during day 6-10 and end of cycle in cycle 1 while on Day 1and end of cycle in subsequent cycles 2 to 6. Summary of mean respiratory rate is presented.
Summary of mean heart rate | Up to end of cycle (approximately 28 days per cycle); maximum up to 24 months
  It was assessed on Day 1, during day 6-10 and end of cycle in cycle 1 while on Day 1and end of cycle in subsequent cycles 2 to 6. Summary of mean heart rate is presented.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (69):
- Argentina (4):
  - GSK Investigational Site, Capital Federal, Buenos Aires
  - GSK Investigational Site, Córdoba, Córdoba Province
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, San Miguel de Tucumán
- Belgium (3):
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Liège
- Bulgaria (2):
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Varna
- GSK Investigational Site, Zagreb, Croatia
- Czechia (5):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Jihlava
  - GSK Investigational Site, Ostrava
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Tábor
- Finland (3):
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Kangasala
  - GSK Investigational Site, Turku
- Greece (4):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Kavala
  - GSK Investigational Site, Papagos, Athens
  - GSK Investigational Site, Thessaloniki
- Hungary (3):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Mátraháza
  - GSK Investigational Site, Székesfehérvár
- India (2):
  - GSK Investigational Site, Kochi
  - GSK Investigational Site, Tirupati
- Ireland (3):
  - GSK Investigational Site, Dublin
  - GSK Investigational Site, Tallaght, Dublin
  - GSK Investigational Site, Wilton, Cork
- Italy (4):
  - GSK Investigational Site, Monteforte Irpino, Campania
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Sassari, Sardinia
  - GSK Investigational Site, Pisa, Tuscany
- Malaysia (3):
  - GSK Investigational Site, George Town
  - GSK Investigational Site, Kubang Kerian
  - GSK Investigational Site, Sarawak
- Pakistan (3):
  - GSK Investigational Site, Islamabad
  - GSK Investigational Site, Karachi
  - GSK Investigational Site, Lahore
- Philippines (3):
  - GSK Investigational Site, Baguio City, Benguet
  - GSK Investigational Site, Manila
  - GSK Investigational Site, Quezon City
- Poland (5):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Olsztyn
  - GSK Investigational Site, Poznan
- Romania (3):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Iași
  - GSK Investigational Site, Timișoara
- Slovakia (3):
  - GSK Investigational Site, Banská Bystrica
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Poprad
- GSK Investigational Site, Seoul, South Korea
- Spain (5):
  - GSK Investigational Site, Ávila
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Murcia
  - GSK Investigational Site, Valencia
- Taiwan (2):
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, TaoYuan Hsien
- Thailand (2):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai
- Ukraine (5):
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Lviv
  - GSK Investigational Site, Sympheropol
  - GSK Investigational Site, Uzhhorod

REFERENCES:
- [Result] Grunberg SM, Rolski J, Strausz J, Aziz Z, Lane S, Russo MW, Wissel P, Guckert M, Wright O, Herrstedt J. Efficacy and safety of casopitant mesylate, a neurokinin 1 (NK1)-receptor antagonist, in prevention of chemotherapy-induced nausea and vomiting in patients receiving cisplatin-based highly emetogenic chemotherapy: a randomised, double-blind, placebo-controlled trial. Lancet Oncol. 2009 Jun;10(6):549-58. doi: 10.1016/S1470-2045(09)70109-3. Epub 2009 May 8. PMID 19428297